CLINICAL TRIAL: NCT06570954
Title: Retraining and Control Therapy (ReACT): Sense of Control and Catastrophic Symptom Expectations as Targets of a Cognitive Behavioral Treatment for Adult Functional Seizures (FS)
Brief Title: Retraining and Control Therapy (ReACT)- Adults
Acronym: ReACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Fobian, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300013382; R61MH127155 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Convulsion, Non-Epileptic
Keywords: ReACT
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Intervention Model Description: Participants 19 years and older with PNES will be prospectively enrolled. Participants will be randomly assigned to one of three conditions: no wait, 3-month waiting period, 6-month waiting period after which they will receive 12 sessions of Retraining and Control Therapy (ReACT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers who conduct baseline and follow-up visits will be blinded to the condition to which the patient has been assigned. The statistician and data manger will be blinded to waiting period the patient got assigned to when analyzing data. The PI and therapists will be blinded to participant's baseline target scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No waiting period (Active Comparator): At the end of the baseline visit, participants will be randomized to receive Retraining and Control Therapy (ReACT) with no waiting period.
  Interventions: Behavioral: ReACT
- 3-month waiting period (Active Comparator): At the end of the baseline visit, participants will be randomized to receive Retraining and Control Therapy (ReACT) after a waiting period of 3 months.
  Interventions: Behavioral: ReACT
- 6-month waiting period (Active Comparator): At the end of the baseline visit, participants will be randomized to receive Retraining and Control Therapy (ReACT) after a waiting period of 6 months.
  Interventions: Behavioral: ReACT

INTERVENTIONS:
Behavioral: ReACT — ReACT is a novel cognitive behavioral treatment and is a PNES intervention that targets sense of control and catastrophic symptom expectations. ReACT consists of 12 sessions of therapy focused on teaching patients to regain control of their body through managing thoughts and behaviors that reinforce the PNES and return to previous activities. The PNES is explained as behaviors learned through classical and operant conditioning.
  Other Names: Retraining and Control Therapy

SUMMARY:
The purpose of this study is to assess sense of control and catastrophic symptom expectations as targets for Retraining and Control Therapy (ReACT- an intervention focused on changing behaviors and thoughts) for treatment of adult psychogenic non-epileptic seizures (PNES, episodes resembling epileptic seizures but with no correlated epileptiform activity). 19 years and older participants diagnosed with PNES who are treated at UAB FND clinic will engage in twelve sessions of ReACT. Participants will be randomly assigned to one of three conditions: no wait, 3-month waiting period, 6-month waiting period. Sense of control over actions will be measured by the magic and turbulence task, a well-validated measure of sense of control. Participants will complete the cold pressor test (CPT) in which participants hold their hand in cool water for as long as possible up to 3 minutes. Catastrophic symptom expectations in response to the CPT will be measured by Pain Catastrophizing Scale (PCS), pain tolerance (time with hand in water) and cortisol response. Target assessments occur 7 days before treatment and 7 days after the 12th treatment session. Participants randomized to the 3-month and 6-month waiting period will also complete these measures one additional time immediately before the beginning of their waiting period. Long term follow-up assessments will occur at 2 months, 6 months and 12 months after the 12th treatment session. PNES frequency will be measured from 30 days before to 12 months after treatment. Participants randomized to the 3-month or 6-month waiting period conditions will log weekly PNES episodes until the start of therapy.

DETAILED DESCRIPTION:
Patients with PNES who are treated at the UAB FND clinic will have the option to complete additional study procedures. Participants will come to our laboratory for a baseline visit and 4 follow-up visits. After the baseline visit, participants are randomly assigned to one of three conditions: no wait, 3-month waiting period, 6-month waiting period. After the assigned waiting period participants will receive 12 sessions of Retraining and Control Therapy (ReACT) as usual in the FND clinic. Therapy sessions are completed via telehealth.

During the baseline visit, participants complete several questionnaires assessing demographics, mood and suicidality, relationships with friends and family, as well as past and current PNES symptoms. They will also complete the childhood trauma questionnaire. The treatment targets (sense of control and catastrophic symptom expectations) are measured by the magic and turbulence computer task and pain tolerance, PCS and cortisol response to the CPT, respectively. PNES diaries are completed to assess PNES frequency over the previous 30 days. Participants randomized to the 3-month or 6-month waiting period conditions will log weekly PNES episodes until the start of therapy. Participants will also complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests. The baseline lab visit lasts about 2.5 hours. Saliva is collected over 1 time point before and 3 time points after the CPT to measure cortisol response to the CPT. Participants also collect 2 saliva samples 24 hours later to serve as a baseline outside of the laboratory setting. Participants will also be given a Respironics Actiwatch Spectrum Pro to track sleep and PNES episode severity and frequency for the 1 week following the baseline visit. Participants randomized to the 3-month and 6-month waiting period will also complete these measures one additional time immediately before the beginning of their waiting period.

After the baseline visit, participants are scheduled for the first of their 12 intervention sessions of ReACT depending on the waiting period they are assigned to. This first session lasts a maximum of two hours, and the following 11 sessions are scheduled weekly and last one hour. All 12 therapy sessions are conducted as telehealth visits via HIPAA-compliant platform. Participants will be mailed another Respironics Actiwatch Spectrum Pro before the 12th therapy session to track sleep and PNES episode severity and frequency for the 1 weeks between the 12th therapy session and the lab visit one week after the 12th treatment session.

Follow-up at 7 days after treatment is conducted to perform tasks and complete follow-up assessment of the targets (sense of control and catastrophic symptom expectations), PNES frequency, and questionnaires. Each of these sessions last 2 hours. Participants will complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests at the lab visit at each of these visits. Participcants will complete 3 follow-up visits via Zoom at 2 months, 6 months and 12 months after treatment to assess long-term PNES outcomes and questionnaire data. These appointments will last 1 hour. PNES frequency will be measured from 30 days before treatment to 12 months after treatment through PNES diaries completed by the participant.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older.
* Diagnosis of psychogenic non-epileptic seizures by a medical doctor using video-EEG.

Exclusion Criteria:

* Comorbid Epilepsy
* Less than 4 PNES per month
* Other paroxysmal nonepileptic events (e.g. episodes related to hypoxic-ischemic phenomena, sleep disorders or migraine-associated disorders)
* Participation in other therapy during the study
* Severe intellectual disability
* Severe mental illness (delusions/hallucinations)

Exclusion for CPT:

• Blood pressure >130/80 mmHg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Magic and turbulence task | 6-12 months
  Measure of perceived sense of control in response to tasks in which control is manipulated; Greater negative numbers indicate improved understanding of control. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Pain catastrophizing scale- situation specific | 6-12 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done after performing Cold Pressor Test. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Pain tolerance (time) | 6-12 months
  Measures catastrophic symptom expectations. Measured by the total time the participant can keep their hand in cool water during the Cold Pressor Test. Shorter time indicates less pain tolerance. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Salivary Cortisol | 6-12 months
  Measures catastrophic symptom expectations. Measured before and after the cold pressor test. Increased cortisol response indicate increased perceived pain severity. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Pain Rating Scale | 6-12 months
  Measures perceived pain severity after the CPT; score ranges from 0-100. Higher scores indicate greater perceived pain severity. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Stroop task | 6-12 months
  Measure of cognitive inhibition and selective attention, higher scores means poorer cognitive inhibition and selective attention. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.

SECONDARY OUTCOMES:
PNES Frequency | 16-22 months
  Measured by Psychogenic Non-epileptic Seizures (PNES) diary, including frequency, premonitory symptoms, description of PNES symptoms and duration. Assessed 30 days before baseline visit to 12 months after the 12th treatment session.
Pain Catastrophizing Scale (PCS)- General | 6-12 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done before performing Cold Pressor Test. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions.
Anxiety Sensitivity Index (ASI) | 16-22 months
  Assesses catastrophic symptom expectations; scores ranges from 0-64, higher scores indicate greater anxiety. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
Shipley | At Baseline
  Assesses verbal IQ; higher scores indicate greater verbal IQ. Completed by participant. Assessed at baseline visit.
Quality of Life in Epilepsy (QOLIE-31) | 16-22 months
  Assesses health-related quality of life for patients with epilepsy (used in PNES participants by instructing them to consider their PNES when asked about "seizures"); score ranges from 0-100, higher scores indicate better functioning and well-being. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions
Sense of Agency Question | 16-22 months
  Single question which asks "How much control do you believe you have over your PNES?", scored using a 4-point Likert scale. Lower score indicates better control over PNES. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
LEVEL 2-Somatic Symptom report adapted from the Participant Health Questionnaire | 16-22 months
  Measures symptom severity; scores ranges from 0-26, higher scores indicate greater symptom severity. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
WHO Disability Assessment Schedule (WHODAS2.0) | 16-22 months
  Completed by participant to measure physical functioning and disability in patients with chronic pain; score ranges from 0-100, higher scores indicate greater perceived functional disability. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions
The Impact on Family Scale | 16-22 months
  Assesses participant's perceptions of the impact of their medical condition on the family; higher scores indicate greater financial burden on the family. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
Childhood Trauma Questionnaire | At baseline
  History of physical, sexual and/or emotional abuse and physical and emotional neglect. All clinical subscales have a score range of 5-25, higher scores indicate greater abuse/neglect. Completed by participant. Assessed at baseline visit.
Hospital Anxiety and Depression Scale (HADS) | 16-22 months
  Measures anxiety and depression symptoms in patients; scores ranges from 0-21 for subscales, higher scores indicate increased symptom severity. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
The Columbia Suicide Severity Rating Scale (C-SSRS) | 16-22 months
  Measure that addresses the full range of suicidal thoughts and behaviors that suggest a person is at heightened risk of committing suicide; score ranges from 0-25, higher score indicates greater suicidal ideation intensity. Completed by trained research study coordinator.Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions.
Healthcare Related Stigma Questionnaire | At baseline
  Measures stigma in patients related to their interaction with health care; scores ranges from 0-64, higher scores indicate greater stigma. Completed by participant. Assessed at baseline visit.
Flanker Inhibitory Control and Attention Subtest | 6-12 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function and attention; higher scores indicate better performance. Completed by participant. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session.
List Sorting Working Memory Subtest | 6-12 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures working memory; higher scores indicate better performance. Completed by participant. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session.
Pattern Comparison Processing Speed Subtest | 6-12 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures processing speed; higher scores indicate better performance. Completed by participant. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session.
Dimensional Change Card Sort Subtest | 6-12 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function; higher scores indicate better performance. Completed by participant. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session.
Picture Sequence Memory Subtest | 6-12 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures episodic memory; higher scores indicate better performance. Completed by participant. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session.
Sleep Duration | 4-10 months
  Measures total sleep duration in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
Sleep Efficiency | 4-10 months
  Measures quality of sleep. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
Sleep Onset Latency | 4-10 months
  Refers to the time it took the child to fall asleep after lying down in bed. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
Sleep - Bed Time | 4-10 months
  Measures total time in bed in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
Sleep - Wake Time | 4-10 months
  Measures total awake time in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
PNES Episode Duration | 4-10 months
  Measures the duration of a PNES episode. Objectively measured using Respironics Actiwatch Spectrum Pro. Worn by participant. Assessed for 1 week between baseline visit and 1st therapy session and 1 week between 12th therapy session and 1 week follow-up visit after treatment.
Rosenberg Self-esteem scale | 16-22 months
  This is a 10-item scale measuring self esteem. Score ranges from 0-30 with low scores indicating low self-esteem. Completed by participant at baseline visit and follow-up visits.
Beaver's Self-Report Family Inventory | At Baseline
  This is a 36 item scale which assesses a family member's view of overall family competence. Completed by participant at baseline visit.
FND Locus of Control: Multidimensional Health Locus of Control (MHLC) Scales | 16-22 months
  Measures an individual's belief in his/her ability to control health outcomes. Form C of MHLC scale will be completed by participant. Assessed at baseline visit and follow-up visits.
Dysfunctional Attitude Scale (DAS-9) | 16-22 months
  Participant will complete this 9-item self-report measure that aims to determine stable negative attitudes that people with depression hold about themselves, the world, and their future. Assessed at baseline visit and follow-up visits.
Mishel Uncertainty in Illness Questionnaire-Community Form (MUIS-C) | 16-22 months
  Participant will complete this 23-item scale which measures uncertainty about their diagnosis. Assessed at baseline visit and follow-up visits.
Revised Helping Alliance Questionnaire- II | 16-22 months
  Revised Helping Alliance Questionnaire-II is a 19-item scale will assess the therapist and participants' perception of the therapeutic alliance at follow-ups. Scores ranges from 19-114 with a higher score indicating better therapeutic alliance. Completed at baseline and follow-up visits.
The Credibility/Expectancy Questionnaire | 16-22 months
  The Credibility/Expectancy Questionnaire will be used to compare treatment expectancy between conditions. It measures how much the patient believes the therapy they are receiving will help to reduce their PNES. This will be completed initially after being randomized, after the first session, 4th session, 8th session and at the follow-up visits.
Session Summary Sheet (SSS) | 6-12 months
  Assesses participant's therapeutic relationship, mastery of skill and involvement in therapy session. Completed by therapist at each intervention visit.
Illness Cognitions Scale | 16-22 months
  Participant will complete this 17-item scale measuring the degree to which they align with the sick role. Assessed at baseline visit and follow-up visits.
Other FND Symptoms Questionnaire | 16-22 months
  Assesses if participant has other functional symptoms (independent from their PNES), and evaluates the intensity and frequency of these symptoms. Completed by parent at Baseline and follow-up visits
Dissociative Experiences Scale | 16-22 months
  Participant assesses this 28 item scale which assesses the severity of dissociation. Score ranges from 0 to 100% with a higher score indication greater dissociation. Completed at baseline and follow-ups.
Life Stress Inventory | 16-22 months
  Participant completes this 43 item scale which assesses susceptability to stress-induced health problems. Scores ranges from 0-430 with a higher score indicating greater susceptability to stress-induced health problems. Completed at baseline and follow-up visits.
Somatoform Dissociative Questionnaire | 16-22 months
  Participant completes this 20 item scale which evaluates the severity of somatoform manifestations of the dissociation of personality. Score ranges from 5-100 and a higher score indicates greater somatoform disorders due to personality dissociation. Completed at baseline and follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fobian, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States